CLINICAL TRIAL: NCT01402076
Title: An Open-Label, Single-Sequence Study to Assess the Effect of Multiple Doses of Tasimelteon on the Cytochrome P450 3A4 and 2C8 Enzymes Using Midazolam and Rosiglitazone as Substrates in Healthy Subjects
Brief Title: A Study to Assess the Effect Tasimelteon on the Cytochrome P450 3A4 and 2C8 Enzymes in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1110
Record Dates: First submitted 2011-07-19; First posted 2011-07-26 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Drug Interaction
MeSH Terms: interventions — tasimelteon; Rosiglitazone; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steady State PK Group (Experimental)
  Interventions: Drug: Tasimelteon; Drug: Rosiglitazone; Drug: Midazolam
- No steady state PK (Experimental)
  Interventions: Drug: Tasimelteon; Drug: Rosiglitazone; Drug: Midazolam

INTERVENTIONS:
Drug: Tasimelteon — 20mg daily dosing, Days 4-20
Drug: Rosiglitazone — 4mg, single dose, Days 3 and 20
  Other Names: Avandia
Drug: Midazolam — 10mg, single dose, Days 1 and 18

SUMMARY:
The purpose of this research study is to understand whether there is any difference in the amount of midazolam (including its breakdown product) in the blood when midazolam is given with tasimelteon, and whether there is any difference in the amount of rosiglitazone in the blood when rosiglitazone is given with tasimelteon.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and acceptance to provide written informed consent;
2. Subjects must be males or females between 18 and 55 years of age, inclusive;
3. Female subjects of childbearing potential must be non-pregnant and non-lactating and have a negative serum or urine pregnancy test at the Screening visit and at Check-in (Days -1) and agree not to attempt to become pregnant during the course of the study. Female subjects of childbearing potential (including peri-menopausal women who have had a menstrual bleeding within 1 year) must be using appropriate birth control (e.g. intrauterine device [IUD], diaphragm or condom with spermicidal jelly or foam or abstinence, or cervical cap) for a period of 35 days before the first dosing, for the duration of the study, and for one month after the last dose;

   a. Note: Women are not permitted to use hormonal methods of birth control (e.g. oral contraceptives, hormonal intrauterine device [IUD], patch and steroids) and must use another acceptable method of birth control during the study and for one month after the last dose. Women currently taking oral contraceptives will be required to discontinue their regimen two weeks prior to first dosing.
4. Subjects with Body Mass Index (BMI) of >18 and <35 kg/m2 (BMI = weight (kg)/ [height (m)]2);
5. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below:

   1. Body temperature between 35.0-37.5 °C;
   2. Systolic blood pressure between 90-150 mm Hg;
   3. Diastolic blood pressure between 50-95 mm Hg;
   4. Pulse rate between 50-100 bpm.
6. Willing and able to comply with study requirements;
7. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis;

Exclusion Criteria:

1. History of recent (within six months) drug or alcohol abuse;
2. Any major surgery within three months of Day 1 or any minor surgery within one month;
3. Donation or loss of 400 mL or more of blood within two months prior to the Baseline Visit;
4. History or current evidence of cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction judged by the Investigator to be clinically significant;
5. Any condition requiring the regular use of medication;
6. History of intolerance and/or hypersensitivity to drugs including midazolam, rosiglitazone or other 'glitazones', melatonin or melatonin agonists, or anyone who has taken a melatonin preparation chronically within the past two months prior to Day 1;
7. History of or current evidence of hypoglycemia judged by the Investigator to be clinically significant;
8. History of liver disease and/or positive for one or more of the following serological results: HCV, HIV, HBsAg
9. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 day preceding Day 1;
10. Elevated (> 2 times the upper limit of normal) liver function tests (i.e. aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), and total bilirubin);
11. Inability to be venipunctured and/or tolerate venous access;
12. Subjects who have used tobacco products 3 months prior to dosing.
13. Exposure to any investigational drug within 30 days or 5 half lives (whichever is longer) of baseline, including placebo;
14. Participation in a previous BMS-214778/VEC-162 trial;
15. Use of prescription or OTC medication, including herbal products (e.g., St. John's Wort) within 2 weeks of Day 1;
16. Use of any food or beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard) and charbroiled meats within 1 week before Day 1 and during the actual duration of the study;
17. Any other sound medical reason as determined by the clinical Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
CYP3A4 Pharmacokinetics | Days 1 and 18
  Composite of 24 hour pharmacokinetic parameters of midazolam will be compared between Day 1 and Day 18.
CYP2C8 Pharmacokinetics | Days 3 and 20
  Composite of 24 hour pharmacokinetic parameters of rosiglitazone will be compared between Day 3 and 20.

SECONDARY OUTCOMES:
Midazolam PK | Days 1 and 17
  Composite pharmacokinetic parameters of midazolam and α-hydroxymidazolam will be compared between Day 1 and Day 18.
Rosiglitazone PK | Days 3 and 20
  Composite of 24 hour pharmacokinetic parameters of rosiglitazone will be compared between Day 3 and Day 20.
Tasimelteon multiple dose pharmacokinetics | Days 4-21
  Composite of 24 hour pharmacokinetic parameters of tasimelteon and tasimelteon metabolites M9, M11, M12, M13, and M14, at Days 5, 8, 11, 14 (Group 1 only), and Days 17 and 19 (Groups 1 and 2).
Tasimelteon safety and tolerability | Days 1-21
  Safety of multiple oral doses of 20 mg of tasimelteon alone and in combination with 10 mg of midazolam as measured by vital signs, ECG, and adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States